CLINICAL TRIAL: NCT03294135
Title: Long Term Immunogenicity up to 15 Years After the First Booster Immunization With GSK Biologicals' Encepur Adults (Polygeline-free Tick-Borne Encephalitis Vaccine for Adults) in Adults Who Received 1 of 3 Different Primary Vaccination Schedules
Brief Title: The Aim of This Study is to Investigate the Persistence of Antibody Response in Adults up to 15 Years After One Booster Dose of GlaxoSmithKline (GSK) Biologicals' Encepur Adults Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205847; 2017-001356-59 (EudraCT Number)
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-09

CONDITIONS: Virus Diseases
Keywords: Encepur; Adults; Long term immunogenicity; Tick-borne Encephalitis vaccine; Booster
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Intervention Model Description: All subjects will come to the yearly scheduled blood draw visit for investigation of 11 to 15 year persistence of Neutralization Test (NT) titres. Subjects who have an NT titre below 10 at one of the scheduled visits will receive a second booster dose 6 months after this visit at an unscheduled visit. Subsequent data of these subjects will be analysed separately in a subgroup.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Group (Experimental): Participants who received primary vaccination in study V48P7 on Days 0, 28 (+10) and 300 (+21) (55 participants) and who received a booster vaccination in study V48P7E1 (NCT00387634) (55 participants). For these participants a second booster vaccination within six months after the annual blood draw was to be administered within the present study only in case their Neutralization Test (NT) titer resulted below 10.
  Interventions: Biological: Encepur Adults
- Accelerated/Rapid Group (Experimental): Participants who received primary vaccination in study V48P7 on Days 0, 7 (+3) and 21 (+7) (66 participants) and who received a booster vaccination either in study V48P7E1 (NCT00387634) (9 participants) or before enrolment in study V48P7E1 (NCT00387634) (40 participants). For these participants a second booster vaccination within six months after the annual blood draw was to be administered within the present study only in case their NT titer resulted below 10.
  Interventions: Biological: Encepur Adults
- Accelerated Conventional Group (Experimental): Participants who received primary vaccination in study V48P7 on Days 0, 14 (+3) and 300 (+21) (133 participants) and who received a booster vaccination in study V48P7E1 (NCT00387634) (109 participants). For these participants a second booster vaccination within six months after the annual blood draw was to be administered within the present study only in case their NT titer resulted below 10.
  Interventions: Biological: Encepur Adults

INTERVENTIONS:
Biological: Encepur Adults — One dose of the vaccine can be administered at any one unscheduled visit depending on the detection of NT below 10. It will be administered intramuscularly into the non-dominant deltoid.

SUMMARY:
The purpose of this study is to continue the evaluation of antibody persistence through 11 to 15 years after first booster with Tick-Borne Encephalitis (TBE) vaccine. This study will further investigate the booster response in subjects who will receive their second booster dose* in this study.

* Any booster given in this study will be the second that the subject has received (with regard to the follow-up of the previous study).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* Subjects who have participated in study V48P7E2 (NCT01562444) and who received in the parent V48P7 study one of the following schedules: rapid, conventional, or accelerated conventional and a booster vaccination in study V48P7E1 (NCT00387634) or before study V48P7E1 (NCT00387634) (only rapid schedule).

Additional inclusion criteria for subjects who will need a second booster dose:

* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female subjects of childbearing potential can receive the booster vaccine in the study, if the subject: has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception for 2 months after booster administration.

Exclusion Criteria:

Each subject must not be:

* Unwilling or unable to give written informed consent to participate in the study.
* Perceived to be unreliable or unavailable to complete the study.

Each subject must not have:

* Clinical conditions representing a contraindication to blood draws.
* Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Levels of NT<10 in V48P7E2 (NCT01562444) study.
* Previous vaccination against TBE or other Flavivirus diseases with other TBE and Flavivirus vaccines (e.g. Yellow fever vaccine, Dengue fever vaccine, Japanese encephalitis vaccine) before, during and after completion of the V48P7E2 (NCT01562444) and before starting TBEV POLYGELINE FREE-025 EXT 21 study.
* Primary immunization with TBE vaccine in the parent study V48P7 according to the modified conventional (MC) schedule.
* History of confirmed TBE infection.
* Known exposure to other Flaviviruses.

Each subject who will receive the second booster vaccination in this study additionally to the exclusion criteria above must not have:

* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination.
* Progressive, unstable or uncontrolled clinical conditions.
* Abnormal function of the immune system resulting from: Clinical conditions. Systemic administration of corticosteroids for more than 14 consecutive days within 90 days prior to informed consent. This will mean prednisone ≥20 mg/day (for adult subjects) or equivalent. Inhaled and topical steroids are allowed. Administration of antineoplastic and immuno-modulating agents or radiotherapy within 90 days prior to vaccination.
* Received immunoglobulins or any blood products within 180 days prior to vaccination.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Acute disease and/or fever at the day of booster vaccination.
* Expected general decrease in immune response.
* Organic brain disturbances, including seizure disorders.
* Progressive neurological disorders.
* Suffered febrile or afebrile convulsions.
* Serious chronic illness.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine or chemically related substances.
* Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to vaccination in this study or who are planning to receive any vaccine within 28 days from the study vaccines.
* Pregnant.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beran J, Lattanzi M, Costantini M, Pammolli A, Galgani I. Sustained antibody persistence for at least 15 years after a booster vaccination against tick-borne encephalitis following different primary vaccination schedules: Third 5-year follow-up. Vaccine. 2023 May 26;41(23):3518-3524. doi: 10.1016/j.vaccine.2023.04.061. Epub 2023 May 3. PMID 37142462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 194 subjects, who participated in study V48P7E2(NCT01562444), received in a parent V48P7 study one of the following primary schedules: rapid(R), conventional(C), or accelerated conventional(AC), who received a booster dose in study V48P7E1(NCT00387634) or before study V48P7E1(only R-schedule), and agreed to participate in this study, were enrolled.
Pre-assignment Details: No participant received vaccination in study V48P7E2 (NCT01562444).
Period: Overall Study
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Started | 50 | 43 | 101
Completed | 46 | 43 | 99
Not Completed | 4 | 0 | 2
Not completed — Serious Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group | Total
Number analyzed (Participants) | 50 | 43 | 101 | 194
Age, Customized [Mean (Standard Deviation); unit: Years] | 47.0 (14.1) | 48.8 (15.3) | 48.1 (14.5) | 48.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 22 | 52 | 105
  Male | 19 | 21 | 49 | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 50 | 43 | 101 | 194

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Detectable TBE Neutralizing Antibody Titers Equal to or Above 10 at Year 11
Description: Antibody titers were measured by GSK Biologicals' Neutralization test. Analysis of the percentages of participants with antibody titers >= 2 was not performed as planned in the protocol, as only 3 participants had antibody titers between 2 and 10 during the whole study period.
Time Frame: At Year 11
Population: The analysis was performed on the Per Protocol set-1 (PPS-1) which consisted of all participants who provided evaluable serum samples at the relevant time points and have no major protocol violation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 48 | 43 | 101
Percentage of participants | 100 [92.6 to 100] | 100 [91.8 to 100] | 99.0 [94.6 to 100]

2. Primary Outcome: Percentage of Participants With Detectable TBE Neutralizing Antibody Titers Equal to or Above 10 at Year 12
Description: as for outcome 1
Time Frame: At Year 12
Population: The analysis was performed on the PPS-1 which consisted of all participants who provided evaluable serum samples at the relevant time points and have no major protocol violation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 50 | 43 | 101
Percentage of participants | 98.0 [89.4 to 99.9] | 100 [91.8 to 100] | 99.0 [94.6 to 100]

3. Primary Outcome: Percentage of Participants With Detectable TBE Neutralizing Antibody Titers Equal to or Above 10 at Year 13
Description: as for outcome 1
Time Frame: At Year 13
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 49 | 43 | 101
Percentage of participants | 95.9 [86.0 to 99.5] | 100 [91.8 to 100] | 99.0 [94.6 to 100]

4. Primary Outcome: Percentage of Participants With Detectable TBE Neutralizing Antibody Titers Equal to or Above 10 at Year 14
Description: as for outcome 1
Time Frame: At Year 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 49 | 43 | 101
Percentage of participants | 95.9 [86.0 to 99.5] | 100 [91.8 to 100] | 99.0 [94.6 to 100]

5. Primary Outcome: Percentage of Participants With Detectable TBE Neutralizing Antibody Titers Equal to or Above 10 at Year 15
Description: as for outcome 1
Time Frame: At Year 15
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 48 | 43 | 100
Percentage of participants | 95.8 [85.7 to 99.5] | 100 [91.8 to 100] | 99.0 [94.6 to 100]

6. Primary Outcome: Geometric Mean Antibody Titers (GMTs) by Age Categories at Year 11
Description: Immunogenicity was measured in terms of GMTs of serum TBE Neutralizing Antibody Titers at Year 11. GMTs were assessed for following age subgroups: 25 to 49 years, equal to or above (>=) 50 years and >= 60 years.
Time Frame: At Year 11
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 48 | 43 | 101
Titers
  25 to 49 Years of Age: number analyzed (Participants) | 24 | 23 | 55
  25 to 49 Years of Age | 368.8 [208.9 to 651.1] | 301.5 [168.7 to 538.7] | 235.2 [161.6 to 342.3]
  >=50 Years of Age: number analyzed (Participants) | 24 | 20 | 46
  >=50 Years of Age | 129.6 [76.7 to 218.8] | 177.4 [100.0 to 314.9] | 128.1 [87.7 to 187.0]
  >=60 Years of Age: number analyzed (Participants) | 12 | 13 | 26
  >=60 Years of Age | 127.5 [61.3 to 265.4] | 160.2 [79.2 to 324.0] | 103.0 [62.6 to 169.5]

7. Primary Outcome: Geometric Mean Antibody Titers (GMTs) by Age Categories at Year 12
Description: Immunogenicity was measured in terms of GMTs of serum TBE Neutralizing Antibody Titers at Year 12. GMTs were assessed for following age subgroups: 25 to 49 years, >= 50 years and >= 60 years.
Time Frame: At Year 12
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 50 | 43 | 101
Titers
  25 to 49 Years of Age: number analyzed (Participants) | 26 | 23 | 55
  25 to 49 Years of Age | 323.7 [185.0 to 566.3] | 334.6 [184.6 to 606.4] | 264.3 [179.9 to 388.3]
  >=50 Years of Age: number analyzed (Participants) | 24 | 20 | 46
  >=50 Years of Age | 154.5 [87.6 to 272.4] | 205.8 [110.6 to 383.0] | 158.2 [105.0 to 238.3]
  >=60 Years of Age: number analyzed (Participants) | 12 | 13 | 26
  >=60 Years of Age | 133.6 [62.5 to 285.6] | 190.8 [92.0 to 395.9] | 141.0 [84.2 to 236.3]

8. Primary Outcome: Geometric Mean Antibody Titers (GMTs) by Age Categories at Year 13
Description: Immunogenicity was measured in terms of GMTs of serum TBE Neutralizing Antibody Titers at Year 13. GMTs were assessed for following age subgroups: 25 to 49 years, >= 50 years and >= 60 years.
Time Frame: At Year 13
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 49 | 43 | 101
Titers
  25 to 49 Years of Age: number analyzed (Participants) | 26 | 23 | 55
  25 to 49 Years of Age | 196.9 [112.2 to 345.6] | 238.4 [131.1 to 433.6] | 172.8 [117.3 to 254.3]
  >=50 Years of Age: number analyzed (Participants) | 23 | 20 | 46
  >=50 Years of Age | 98.3 [56.6 to 170.9] | 132.1 [73.0 to 238.9] | 110.9 [75.0 to 164.0]
  >=60 Years of Age: number analyzed (Participants) | 12 | 13 | 26
  >=60 Years of Age | 93.5 [44.7 to 195.6] | 114.8 [56.5 to 233.4] | 96.9 [58.7 to 160.0]

9. Primary Outcome: Geometric Mean Antibody Titers (GMTs) by Age Categories at Year 14
Description: Immunogenicity was measured in terms of GMTs of serum TBE Neutralizing Antibody Titers at Year 14. GMTs were assessed for following age subgroups: 25 to 49 years, >= 50 years and >= 60 years.
Time Frame: At Year 14
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 49 | 43 | 101
Titers
  25 to 49 Years of Age: number analyzed (Participants) | 26 | 23 | 55
  25 to 49 Years of Age | 299.7 [164.2 to 547.0] | 299.1 [157.8 to 567.1] | 248.2 [164.1 to 375.4]
  >=50 Years of Age: number analyzed (Participants) | 23 | 20 | 46
  >=50 Years of Age | 147.5 [81.2 to 268.0] | 169.7 [89.5 to 321.8] | 131.1 [86.0 to 200.0]
  >=60 Years of Age: number analyzed (Participants) | 12 | 13 | 26
  >=60 Years of Age | 139.4 [67.2 to 289.3] | 149.9 [74.3 to 302.4] | 117.9 [71.8 to 193.7]

10. Primary Outcome: Geometric Mean Antibody Titers (GMTs) by Age Categories at Year 15
Description: Immunogenicity was measured in terms of GMTs of serum TBE Neutralizing Antibody Titers at Year 15. GMTs were assessed for following age subgroups: 25 to 49 years, >= 50 years and >= 60 years.
Time Frame: At Year 15
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 48 | 43 | 100
Titers
  25 to 49 Years of Age: number analyzed (Participants) | 26 | 23 | 55
  25 to 49 Years of Age | 217.6 [125.2 to 378.2] | 281.6 [156.5 to 506.9] | 183.9 [125.7 to 268.9]
  >=50 Years of Age: number analyzed (Participants) | 22 | 20 | 45
  >=50 Years of Age | 98.9 [54.4 to 180.0] | 157.0 [83.8 to 294.1] | 103.3 [67.9 to 156.9]
  >=60 Years of Age: number analyzed (Participants) | 11 | 13 | 25
  >=60 Years of Age | 114.1 [52.5 to 247.8] | 158.1 [77.5 to 322.7] | 90.7 [54.2 to 151.7]

11. Secondary Outcome: Percentage of Participants With Detectable TBE Neutralizing Antibody Titers Equal to or Above 2 and Equal to or Above 10 as Measured by GSK Biologicals' NT, Overall and by Study Group
Description: Immunogenicity was planned to be measured in terms of percentage of participants with TBE Neutralizing Antibody Titers >= 2 and >= 10 at 21 days after the booster vaccination.
Time Frame: At 21 days after the booster vaccination
Population: The analysis was planned to be performed on the PPS-2 which consisted of all participants who provided evaluable serum samples after booster dose and have no major protocol violation. However only 1 participant received the booster dose, therefore the analysis was not performed.
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Geometric Mean Antibody Titers (GMTs) as Measured by GSK Biologicals' NT, Overall and by Study Group
Description: Immunogenicity was planned to be measured in terms of GMTs of serum TBE Neutralizing Antibody Titers at 21 days after the booster vaccination.
Time Frame: At 21 days after the booster vaccination
Population: The analysis was planned to be performed on the PPS-2 which consisted of all subjects who provided evaluable serum samples after booster dose and have no major protocol violation. However only 1 participant received the booster dose, therefore the analysis was not performed.
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Geometric Mean Ratios (GMRs) Blood Draw After/Before Booster as Measured by GSK Biologicals' NT, Overall and by Study Group
Description: Immunogenicity was planned to be measured in terms of GMRs of serum TBE Neutralizing Antibody Titers at 21 days after the booster vaccination.
Time Frame: At 21 days after the booster vaccination
Population: as for outcome 12
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants With Detectable TBE Neutralizing Antibody Titers Equal to and Above 10 as Measured by GSK Biologicals' NT, Overall and by Study Group
Description: Immunogenicity was measured in terms of percentage of participants with TBE Neutralizing Antibody Titers >= 10 from Year 1 to Year 15.
Time Frame: From Year 1 up to Year 15
Population: The analysis was performed on the set of subjects who completed the entire 15-year follow-up with no protocol deviations related to the persistence analysis. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
Number analyzed (Participants) | 48 | 43 | 100
Percentage of participants
  Year 1: number analyzed (Participants) | 47 | 42 | 100
  Year 1 | 100 [92.5 to 100] | 100 [91.6 to 100] | 100 [96.4 to 100]
  Year 2: number analyzed (Participants) | 48 | 42 | 99
  Year 2 | 100 [92.6 to 100] | 100 [91.6 to 100] | 100 [96.3 to 100]
  Year 3: number analyzed (Participants) | 48 | 42 | 100
  Year 3 | 100 [92.6 to 100] | 100 [91.6 to 100] | 100 [96.4 to 100]
  Year 4: number analyzed (Participants) | 46 | 41 | 100
  Year 4 | 100 [92.3 to 100] | 97.6 [87.1 to 99.9] | 100 [96.4 to 100]
  Year 5 | 100 [92.6 to 100] | 100 [91.8 to 100] | 100 [96.4 to 100]
  Year 6 | 100 [92.6 to 100] | 100 [91.8 to 100] | 100 [96.4 to 100]
  Year 7: number analyzed (Participants) | 48 | 43 | 98
  Year 7 | 100 [92.6 to 100] | 100 [91.8 to 100] | 100 [96.3 to 100]
  Year 8: number analyzed (Participants) | 47 | 42 | 97
  Year 8 | 100 [92.5 to 100] | 100 [91.6 to 100] | 100 [96.3 to 100]
  Year 9: number analyzed (Participants) | 45 | 42 | 97
  Year 9 | 100 [92.1 to 100] | 100 [91.6 to 100] | 100 [96.3 to 100]
  Year 10: number analyzed (Participants) | 46 | 42 | 98
  Year 10 | 100 [92.3 to 100] | 100 [91.6 to 100] | 100 [96.3 to 100]
  Year 11: number analyzed (Participants) | 46 | 43 | 100
  Year 11 | 100 [92.3 to 100] | 100 [91.8 to 100] | 99.0 [94.6 to 100]
  Year 12 | 97.9 [88.9 to 99.9] | 100 [91.8 to 100] | 99.0 [94.6 to 100]
  Year 13 | 95.8 [85.7 to 99.5] | 100 [91.8 to 100] | 99.0 [94.6 to 100]
  Year 14 | 95.8 [85.7 to 99.5] | 100 [91.8 to 100] | 99.0 [94.6 to 100]
  Year 15 | 95.8 [85.7 to 99.5] | 100 [91.8 to 100] | 99.0 [94.6 to 100]

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs are defined as any untoward medical occurrence that results in death, is life- threatening, requires hospitalisation or prolongation of existing hospitalisation, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to Day 21 after booster vaccination
Population: The analysis was performed on the Safety population which included all subjects who received a booster vaccination in this study. Only one participant (from the Conventional Group) received a booster dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Group
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events that led to withdrawal or were related to study vaccination were collected throughout the study period (Year 11 to Year 15). Other serious adverse events were collected only after the booster vaccination administration (Day 0-Day 21).
Description: Other adverse events were not collected as per protocol.
Arm/Group | Conventional Group | Accelerated/Rapid Group | Accelerated Conventional Group
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/43 | 1/101
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/43 | 1/101
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Group (N=50) | Accelerated/Rapid Group (N=43) | Accelerated Conventional Group (N=101)
Death due to glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Death due to primary COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT03294135/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT03294135/SAP_001.pdf